CLINICAL TRIAL: NCT03179605
Title: An Open Label, Multicenter Study to Assess the Potential for Adrenal Suppression and Systemic Drug Absorption Following Multiple Dosing With DFD-06 in Pediatric Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: Assess the Potential for Adrenal Suppression and Systemic Drug Absorption Following Multiple Dosing With DFD-06
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty in enrollment
Sponsor: Primus Pharmaceuticals (Industry)
Collaborators: Prosoft Clinical (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DFD-06-CD-011
Record Dates: First submitted 2017-05-12; First posted 2017-06-07 (Actual); Results first posted 2022-06-01 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Clobetasol

STUDY DESIGN:
Intervention Model Description: In the first stage, subjects who are at least 12 years of age and not more than 16.9 years (16 years and 11 months) of age with moderate to severe plaque psoriasis will be treated with DFD-06 (at least 20 completed subjects). In the second stage subjects who are at least 6 years of age and not more than 11.9 years (11 years and 11 months) of age with moderate to severe plaque psoriasis will be treated with DFD-06 (at least 20 completed subjects).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DFD-06 Cream (Experimental): This is a single arm, open label study and there will be no reference or control product used in this study
  Interventions: Drug: DFD06

INTERVENTIONS:
Drug: DFD06 — Apply twice per day for 15 days
  Other Names: clobetasol propionate, Impoyz Cream

SUMMARY:
The purpose of this study is to evaluate the potential of DFD-06 to suppress the hypothalamic-pituitary-adrenal (HPA) axis when applied twice daily for 15 days.

DETAILED DESCRIPTION:
This is a 15-day, single arm, multicenter, multi-dose, open-label, two stage, sequential study. In the first stage, subjects who are at least 12 years of age and not more than 16.9 years (16 years and 11 months) of age with moderate to severe plaque psoriasis will be treated with DFD-06 (at least 20 completed subjects). In the second stage subjects who are at least 6 years of age and not more than 11.9 years (11 years and 11 months) of age with moderate to severe plaque psoriasis will be treated with DFD-06 (at least 20 completed subjects). An attempt will be made to enroll subjects throughout the age range of each cohort including the lower age range. DFD-06 will be applied twice daily to all affected areas on the body excluding face, scalp, groin, axillae and other intertriginous areas. Subjects must have ≥10% Body Surface Area (BSA) treated to achieve maximal use exposure.

ELIGIBILITY:
Inclusion Criteria:

* Subjects and the parent or legal guardian understand the study procedures and agree to participate by giving assent and written informed consent, respectively. Subject's parent or legal guardian must be willing to authorize use and disclosure of protected health information collected for the study.
* Subjects must be at least 6 years and not more than 16.9 years of age, with body weight greater than or equal to 45 pounds at Screening.
* Subjects must present with a clinical diagnosis of stable (at least 3 months) plaque psoriasis.
* Subjects with psoriasis involving ≥10% Body Surface Area (BSA), not including the face, scalp, groin, axillae and other intertriginous areas at the Baseline Visit.
* Subjects must have an Investigator Global Assessment (IGA) grade of at least 3 (moderate) at the Baseline Visit.

Exclusion Criteria:

* Subject has a current diagnosis of unstable forms of psoriasis including guttate, erythrodermic, exfoliative or pustular psoriasis.
* Subject has a history of organ transplant requiring immunosuppression, HIV, or other immunocompromised state.
* Subject has received treatment for any type of cancer within 5 years of the Baseline Visit except skin cancer and cervical cancer (in situ) are allowed if at least 1 year before the Baseline Visit.
* Subject has a history or presence of intracranial hypertension.
* Subject has had prolonged exposure to natural or artificial sources of ultraviolet radiation within 30 days prior to the initiation of treatment or is intending to have such exposure during the study that is thought by the investigator to likely modify the subject's disease

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2019-06-03 (Actual); Study Completion 2020-06-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Site 104, Madera, California
  - Site 108, Santa Ana, California
  - Investigational Site 102, Hialeah, Florida
  - Site 109, Hialeah, Florida
  - Site 107, Overland Park, Kansas
  - Site 103, St Louis, Missouri
  - Investigational Site 101, Lincoln, Nebraska
  - Site 106, Greenville, South Carolina
  - Site 105, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Normal response to cosyntropin stimulation defined as a Screening Cosyntropin Stimulation Test (CST) with a 30-minute post-stimulation cortisol level of > 18 ug/dL.
Period: Overall Study
Arm/Group | DFD-06 Cream
Started | 22
Completed | 21
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | DFD-06 Cream
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.2 (1.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 5
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 22
Investigator Global Assessment [Mean (Standard Deviation); unit: units on a scale] — Investigator Global Assessment of psoriasis on a scale of 0 to 5. 0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe
  units on a scale | 3 (0)
Percent Body Surface Area Affected [Mean (Full Range); unit: percent body surface area] — Psoriasis >= 10% body surface area required for enrollment
  percent body surface area | 14.2 [10 to 24]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With HPA Axis Suppression at Day 15
Description: The percentage of subjects with abnormal cortisol response for ACTH stimulation test at Day 15 (cortisol level ≤18 µg/dL at 30 minutes post stimulation) is the primary variable
Time Frame: Day 15
Population: The Evaluable population included those subjects in the Safety population who had both Screening and Day 15 serum cortisol data (pre- and post-cosyntropin stimulation) and had a normal response to Screening Cosyntropin Stimulation Test with a 30-minute post-stimulation cortisol level of > 18 μg/dL and applied at least 80% of expected (29) applications
Measure: Count of Participants; unit: Participants
Arm/Group | DFD-06 Cream
Number analyzed (Participants) | 21
Participants | 3

2. Secondary Outcome: Number of Participants With Improvement in IGA Grade From Baseline
Description: Numbers of subjects with improvements by at least 1 pint in IGA grade will be provided as descriptive statistics.
Time Frame: Baseline up to Day 15
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | DFD-06 Cream
Number analyzed (Participants) | 21
participants
  Day 8 1-point improvement in IGA | 15
  Day 8 2-point improvement in IGA | 2
  Day 15 1 point improvement in IGA | 8
  Day 15 2-point improvement in IGA | 10
  Day 15 3-point improvement in IGA | 2

3. Secondary Outcome: Plasma Concentration of Clobetasol Propionate
Description: Plasma concentrations of clobetasol propionate after multiple doses of DFD-06 under maximal use condition with the final-to-be-marketed formulation.
Time Frame: Day 15 0 hour, 1 hour, 3 hours, 6 hours after application
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | DFD-06 Cream
Number analyzed (Participants) | 8
pg/mL
  0 hour clobetasol plasma level: number analyzed (Participants) | 7
  0 hour clobetasol plasma level | 51.486 (48.35)
  1 hour clobetasol plasma level | 40.370 (32.55)
  3 hour clobetasol plasma level: number analyzed (Participants) | 7
  3 hour clobetasol plasma level | 64.250 (41.93)
  6 hour clobetasol plasma level: number analyzed (Participants) | 7
  6 hour clobetasol plasma level | 42.143 (27.32)
  Average of 1, 3 and 6 hour | 45.47 (32.49)

ADVERSE EVENTS:
Time Frame: 1 month
Description: Adverse events were collected at every visit (except Screening) by spontaneous reports from subjects and legal guardian, either verbal or recorded in the subject diary, by directed questioning of subjects and legal guardian, and by observation.
Arm/Group | DFD-06 Cream
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 8/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DFD-06 Cream (N=22)
HPA Axis Suppression (Endocrine disorders) | 3 (3)
Application Site Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Application Site Pain (Skin and subcutaneous tissue disorders) | 1 (1)
Vein collapse (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination due to low enrollment with completion of 12 to 16.9 years old group only; the planned 6 to 11.9 years of age did not enroll.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-26): https://cdn.clinicaltrials.gov/large-docs/05/NCT03179605/Prot_SAP_001.pdf